CLINICAL TRIAL: NCT06437158
Title: Efficacy and Safety of Different Concentrations of Bleomycin in the Sclerotherapy of Lymphatic Malformations for Pediatric Patients
Brief Title: Use of Bleomycin in the Sclerotherapy of Lymphatic Malformations for Pediatric Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yi Ji, Clinical Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-12-19
Record Dates: First submitted 2023-12-19; First posted 2024-05-31 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Lymphatic Malformation
Keywords: Lymphatic Malformation; Bleomycin; Sclerotherapy; Intracystic injection; High-dose concentrations; Low-dose concentrations
MeSH Terms: conditions — Lymphatic Abnormalities | interventions — Bleomycin; Zeocin

STUDY DESIGN:
Intervention Model Description: The investigators aim to compare the efficacy and safety of different concentrations of Bleomycin in the sclerotherapy of lymphatic malformations for pediatric patients.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-dose Concentrations (1mg/ml) of Bleomycin (Experimental): In this arm, patients with lymphatic malformations were treated by intracapsular injection with low-dose concentrations (1mg/ml) of Bleomycin.
  Interventions: Drug: Bleomycin
- High-dose Concentrations (2mg/ml) of Bleomycin (Experimental): In this arm, patients with lymphatic malformations were treated by intracapsular injection with high-dose concentrations (2mg/ml) of Bleomycin.
  Interventions: Drug: Bleomycin

INTERVENTIONS:
Drug: Bleomycin — To validated the efficacy and safety of different concentrations of Bleomycin in the sclerotherapy of lymphatic malformations for pediatric patients
  Other Names: Zeocin

SUMMARY:
Bleomycin has nowadays been more and more widely used in the sclerotherapy of LMs, which has been proven to be primarily dose dependent. The investigators aim to compare the efficacy and safety of different concentrations of Bleomycin in the sclerotherapy of LMs for pediatric patients.

DETAILED DESCRIPTION:
Lymphatic malformations (LMs) are vascular anomalies that arise from abnormal embryonic development of the lymphatic system and might present as dilated lymphatic channels or cysts lined by lymphatic endothelial cells. With an estimated incidence of approximately 1/4000-1/2000, LMs can occur at any site in the lymphatic system, in which head, neck and axilla were mostly detected and have been reported to account for over 75%. Based on the location and size of the lesion and the extent of involvement, LMs may be asymptomatic with incidental detection, or chronic abdominal pain and distension due to their compression of surrounding structures, or critical and even fatal secondary to their volvulus, hemorrhage, infection and rupture. Surgical excision is a definitive treatment for LMs, while it may be difficult at times because of the infiltrative nature of the lesions, leading to a high incidence of complications like vital organ injuries, nerve injuries, bleeding, infection scar formation, and recurrences. Sclerotherapy is a simpler alternative to tedious surgical excision treatment for LMs and avoids the complications related to surgery. As an anticancer drug extracted from Streptomyces verticillus, Bleomycin has been more and more widely used in the sclerotherapy of LMs for pediatric patients, which has been proven to be primarily dose dependent. However, the optimum concentration of Bleomycin in the sclerotherapy of LMs for pediatric patients has not been strictly validated, due to the lack of high-quality RCT studies. The investigators aim to compare the efficacy and safety of different concentrations of Bleomycin in the sclerotherapy of LMs for pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants less than 14 years of age at the time of informed consent/assent form was signed.
* Participants whose parents have voluntarily given written consent and participants who provided assent (if applicable) after the study has been explained to them.
* Participants with LMs of all sites measured and confirmed via imaging at screening, with rapid progression, resluting in obvious symptoms or dysfunction, which could not be radically resected and could be treated by sclerotherapy.

Exclusion Criteria:

* Penicillin allergy.
* Vascular tumors or combined vascular malformations.
* Participants who may have had surgical or sclerotherapy treatment by other hardeners.
* LMs growing slowly, without obvious symptoms or dysfunction, which does not need to be treated prematurely.

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of Volume | 3 to 6 months post-therapy
  Changes of Volume is defined as follows: a complete (90%-100% reduction in LMs volume), substantial (60%-89% reduction in LMs volume), intermediate (20%-59% reduction in LMs volume), or no (< 20% reduction in LMs volume) response 3 to 6 months post-therapy as assessed by imaging.

SECONDARY OUTCOMES:
Score of Pain | 3 to 6 months post-therapy
  Score of Pain is selfassessed at each visit on a 0 to 10 visual analog scale (where 0 indicates no pain and 10 indicates the worst pain imaginable), reported along with period duration.
Global Efficacy | 3 to 6 months post-therapy
  Global efficacy is assessed at each visit beginning at MS by the physician and self-assessed by the participant and proxy (parents) on a 0 to 10 visual analog scale (where 0 indicates no efficacy and 10 indicates complete resolution).
Score of Quality of Life | 3 to 6 months post-therapy
  Score of Quality of Life is assessed by the validated Children-Dermatological Life Quality Index (C-DLQI).
Number of Participants with Efficacy | 3 to 6 months post-therapy
  Number of Participants with Efficacy was assessed by 2 independent experts.
Number of Participants with Safety | 3 to 6 months post-therapy
  Number of Participants with Safety was assessed based on physical signs and monitoring of imaging examinations or laboratory test.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sun J, Wang C, Li J, Song D, Guo L. The efficacy of bleomycin sclerotherapy in the treatment of lymphatic malformations: a review and meta-analysis. Braz J Otorhinolaryngol. 2023 Jul-Aug;89(4):101285. doi: 10.1016/j.bjorl.2023.101285. Epub 2023 Jun 29. PMID 37423005
- [Result] De Maria L, De Sanctis P, Balakrishnan K, Tollefson M, Brinjikji W. Sclerotherapy for lymphatic malformations of head and neck: Systematic review and meta-analysis. J Vasc Surg Venous Lymphat Disord. 2020 Jan;8(1):154-164. doi: 10.1016/j.jvsv.2019.09.007. Epub 2019 Nov 14. PMID 31734224
- [Result] Wu Z, Zou Y, Fu R, Jin P, Yuan H. A nomogram for predicting sclerotherapy response for treatment of lymphatic malformations in children. Eur J Med Res. 2022 Oct 21;27(1):209. doi: 10.1186/s40001-022-00844-3. PMID 36271467